CLINICAL TRIAL: NCT01750801
Title: Clinical Evidence Efficacy of a Mouthwash Containing Propolis for the Control of Plaque and Gingivitis: Phase III, Randomized, Double-blind Comparison With Mouthwash Chlorhexidine Base.
Brief Title: Efficacy of a Mouthwash Containing Propolis
Acronym: PRO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Andre Oliveira Naufel de Toledo, Principal Investigator, Federal University of Minas Gerais
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Propolis
Record Dates: First submitted 2012-11-22; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Gingivitis; Periodontitis; Plaque; Inflammation
Keywords: clinical trial; mouthwash; propolis; plaque; gingivitis; compliance
MeSH Terms: conditions — Gingivitis; Periodontitis; Plaque, Amyloid; Inflammation; Patient Compliance | interventions — Propolis; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propolis (Active Comparator): alcohol-free mouthwash containing 5% green propolis (MGP 5%) on the control of plaque and gingivitis.
  Interventions: Drug: chlorhexidine
- chlorhexidine (Active Comparator): chlorhexidine used on the control of plaque and gingivitis.
  Interventions: Drug: Propolis

INTERVENTIONS:
Drug: Propolis — Twenty-five subjects, both male and female, were chosen after signing the terms of agreement.. The criteria for selection stated that subjects should be from 18 to 60 years old, should present good health, a minimum of 20 teeth and not be pregnant or breastfeeding.The subjects went through a dental prophylaxis before starting rinse. They were then instructed to rinse twice a day for a minute, immediately after brushing (morning and night), using the 10 ml of the MGP 5%. After 45 and 90 days using the product the individuals returned for a clinical evaluation which considered changes in the soft and hard oral tissues and involved collecting plaque and gingivitis indexes. On their last appointment the subjects answered a questionnaire about their level of appreciation and acceptability of the mouthwash
  Arms: chlorhexidine
Drug: chlorhexidine — Twenty-five subjects, both male and female, were chosen after signing the terms of agreement.The subjects went through a dental prophylaxis before starting rinse. They were then instructed to rinse twice a day for a minute, immediately after brushing (morning and night), using the 10 ml of the MGP 5%. After 45 and 90 days using the product the individuals returned for a clinical evaluation which considered changes in the soft and hard oral tissues and involved collecting plaque and gingivitis indexes. On their last appointment the subjects answered a questionnaire about their level of appreciation and acceptability of the mouthwash
  Arms: Propolis

SUMMARY:
Characterization of green propolis and development of mouthwash containing propolis to control plaque and gingivitis. A Phase I.

DETAILED DESCRIPTION:
Chemical characterization of propolis by HPLC (High-performance liquid chromatography), antimicrobial testing against pathogens and cariogenic. Studies in vitro on anti-inflammatory activity, cytotoxicity tests of green propolis.

ELIGIBILITY:
Inclusion Criteria:

* age ranging from 18 to 60 years
* minimum of 20 natural teeth
* mean plaque index (PI)of at least 1.5
* an average gingival index (GI), at least less than 1.0.

Exclusion Criteria:

* Individuals with orthodontic appliances or removable dentures,
* Individuals whit tumors of soft tissue or hard mouth, and advanced periodontal disease,
* Indivuduals whit antibiotic therapy 2 weeks prior to study initiation, or with known hypersensitivity propolis are also excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Chemical characterization of propolis by HPLC (High-performance liquid chromatography) | 8-12 weeks

SECONDARY OUTCOMES:
PRELIMINARY EVIDENCE OF THE EFFICACY OF A MOUTHWASH CONTAINING 5% PROPOLIS FOR THE CONTROL OF PLAQUE AND GINGIVITIS | 90 days
  After 45 and 90 days using Propolis or chlorhexidine at home, the individuals will return for a clinical evaluation. Alterations in gingival conditions will be analyzed ,both points of comparison products will be based on the Plaque Index of Quigley-Hein and modified gingival index of Loe-Silness modified as scores for the corresponding gravity, being a non-parametric distribution, will be compared by analysis of covariance, by Friedman test for those data to be obtained and analysed the use efficacy after 45 and 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: andre oliveira naufel de toledo 35893/MG, Principal Investigator — UFMG
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil